CLINICAL TRIAL: NCT03733756
Title: to Explore the Influence of Longitudinal Muscle on the Prognosis of Achalasia Patients After Peroral Endoscopic Myotomy
Brief Title: to Explore the Influence of Longitudinal Muscle on the Prognosis of Achalasia Patients After Peroral Endoscopic Myotomy (POEM)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: LM for achalasia
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Esophageal Achalasia
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POEM preserving longitudinal muscle (Experimental): participants are operated POEM only involving circular muscle, leaving longitudinal muscle intact
  Interventions: Procedure: POEM preserving longitudinal muscle
- POEM involving longitudinal muscle (Active Comparator): participants are operated POEM involving the whole layer of muscle, both circular and longitudinal muscle
  Interventions: Procedure: POEM involving longitudinal muscle

INTERVENTIONS:
Procedure: POEM preserving longitudinal muscle — participants are operated POEM only involving circular muscle, leaving longitudinal muscle intact
  Arms: POEM preserving longitudinal muscle
Procedure: POEM involving longitudinal muscle — participants are operated POEM involving both circular and longitudinal muscle
  Arms: POEM involving longitudinal muscle

SUMMARY:
Achalasia is a disease characterized by lack of peristalsis and lower esophageal sphincter failing to relax. Longitudinal muscle, outer layer of esophageal smooth muscle, is recently found to be responsible for emptying of esophagus for achalasia patients, especially for those type Ⅱcases. Clinical observations also conclude that type Ⅱ achalasia which still preserve longitudinal muscle response best to treatment, among the 3 types. Thus, with high frequent intraluminal ultrasound, clinically applied as endoscopic ultrasound, to measure the function of longitudinal muscle in achalasia patients, the current research aims to explore the influence of longitudinal muscle on the prognosis of achalasia patients after peroral endoscopic myotomy, a routine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed of esophageal achalasia
* Patients or legal surrogates willing and competent to give informed consent

Exclusion Criteria:

* postoperative or post-POEM
* post-pneumatic dilation or post-stenting
* fail to go through high frequency intraluminal ultrasound （HFIUS)
* Patients with American Society of Anesthesiologists （ASA） score ≥3

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 308 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
efficacy of POEM treatment | 4 weeks after POEM
  Eckardt score ≤3; Eckardt scale includes 4 items: dysphagia, weight loss, poststernal pain and esophageal reflux, each item ranging from 0-3. The higher the score reaches, the more severe the disease is. It is considered to be efficient if the Eckardt score is ≤3 after POEM.

SECONDARY OUTCOMES:
complications(GERD) of POEM treatment | 4 weeks after POEM
  gastroesophageal reflux disease questionnaire （GERD-Q） score≥2; GERD-Q scale includes 4 items: post-sternal pain, esophageal reflux, proton pump inhibitor applied, endoscopy identified, each item scoring 0 or 1. The higher the score reaches, the more likely the patient has GERD. It is considered to have a complication as GERD if the GERD-Q ≥2.

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Hong Zhou, MD,PhD, Study Chair — Zhongshan Hospital, Fudan University, Shanghai, China
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hong SJ, Bhargava V, Jiang Y, Denboer D, Mittal RK. A unique esophageal motor pattern that involves longitudinal muscles is responsible for emptying in achalasia esophagus. Gastroenterology. 2010 Jul;139(1):102-11. doi: 10.1053/j.gastro.2010.03.058. Epub 2010 Apr 8. PMID 20381493
- [Background] Schoeman MN, Holloway RH. Secondary oesophageal peristalsis in patients with non-obstructive dysphagia. Gut. 1994 Nov;35(11):1523-8. doi: 10.1136/gut.35.11.1523. PMID 7828966
- [Background] Liu ZQ, Li QL, Chen WF, Zhang XC, Wu QN, Cai MY, Qin WZ, Hu JW, Zhang YQ, Xu MD, Yao LQ, Zhou PH. The effect of prior treatment on clinical outcomes in patients with achalasia undergoing peroral endoscopic myotomy. Endoscopy. 2019 Apr;51(4):307-316. doi: 10.1055/a-0658-5783. Epub 2018 Sep 27. PMID 30261536
- [Background] Mittal RK, Liu J, Puckett JL, Bhalla V, Bhargava V, Tipnis N, Kassab G. Sensory and motor function of the esophagus: lessons from ultrasound imaging. Gastroenterology. 2005 Feb;128(2):487-97. doi: 10.1053/j.gastro.2004.08.004. PMID 15685559